CLINICAL TRIAL: NCT04219072
Title: Clinical Classification of Pain in Breast Cancer Survivors: Nociceptive, Neuropathic or Nociplastic Pain
Brief Title: Clinical Classification of Pain in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: KutahyaMSUcancer
Record Dates: First submitted 2019-12-25; First posted 2020-01-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Cancer Pain; Breast Cancer
MeSH Terms: conditions — Chronic Pain; Cancer Pain; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Breast cancer is the most common malignancy in women worldwide according to International Agency for Research on Cancer. Unfortunately, cancer survivors often face long-term symptoms that occur or persist after completion of treatment. In addition to fatigue, pain is the most common persistent symptom after cancer and cancer treatment. The diagnosis and treatment of pain in cancer survivors is not clear for many physicians. A mechanism-based classification of pain in cancer survivors might be a critical step for clinical reasoning, especially for discrimination of different pain types. The primary aim of this study is to determine the prevalence of the predominant type of pain in Turkish breast cancer survivors using a recent published clinical algorithm.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with histologically confirmed invasive or non-invasive primary breast cancer
* completed remission and their primary treatment at least 3 months prior to study participation
* experienced pain or a sensitive disorder (like numbness, tingling, etc.) anywhere in body for which they stated a minimum score of 3 on a numeric pain rating scale

Exclusion Criteria:

* patients affected by other chronic disease,
* severe psychological disorders
* active metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The convenience sampling will implement for this cross-sectional study. Breast cancer survivors experiencing chronic pain who presented at the Department of Oncology of Kutahya Health Sciences University Evliya Celebi Hospital will screen for eligibility by their physician and were subsequently requested to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 1 minute
  The NPRS was used to assess the participants' pain levels. In the NPRS, patients are asked to verbally rate the severity of their pain on a scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Margolis Pain Diagram | 5 minute
  The Margolis Pain Diagram, consists of a dorsal and a ventral drawing body, is used to assess the location and distribution of the pain. Participants will ask to point out the place where they experience pain during the preceding 4 weeks for at least 24 hours
Central Sensitization Inventory | 10 minute
  The Central Sensitization Inventory (CSI) aims to evaluate symptoms thought to be associated with nociplastic pain. The CSI consists 25 items exploring emotional and somatic disorders associated with CS. Each response is scored from 0 to 4, yielding a total score of 0 to 100. A score of 40 or higher on the CSI means the presence of nociplastic pain.
Short Form 36 | 10 minute
  The Short Form-36 (SF-36) is widely used to measurement of health related quality of life (HRQoL) questionnaire. SF-36 is a 36-item generic self-administered instrument consisting of 8 subscales related to various aspects of HRQoL: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The 8 subscales are scored from 0 to 100, with higher scores indicating better health status.

SECONDARY OUTCOMES:
Quantitative sensory test | 10 minute
  Quantitative sensory testing (QST) is a psychophysical method used to quantify somatosensory function in patients. In QST will be used various stimuli static thermal (thermotest), static mechanical ( a painter brush), pinprick (a calibrated pin) and vibration ( a tuning folk). QST will interrogate whether each stimulus is considered a sensory loss (negative sign) or sensory gain (positive sign or hyperalgesia).

CONTACTS AND LOCATIONS:
Locations (1):
- KutahyaMSU, Kütahya, Kutahya Health Sciences University, Turkey (Türkiye)